CLINICAL TRIAL: NCT04641039
Title: Effect of the Postoperative Prevertebral Scar on Controlling Excess After Removing the Anterior Lumbar Disc Annulus Fibrosus to Implant a Lumbar Disc Prosthesis. Biomechanical and Clinical Study
Brief Title: Postoperative Scar in the Control Excess of Mobility Induced by Annulus Removal on Inserting a Lumbar Disc Prosthesis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, Vicente Vanaclocha, Profesor of Neurosurgery, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 101/2020
Record Dates: First submitted 2020-11-12; First posted 2020-11-23 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Lumbar Disc Disease
Keywords: Annulus fibrosus; Lumbar disc prosthesis; Lumbar disc replacement; Range of movement lumbar disc prosthesis; Quality of life after lumbar disc replacement
MeSH Terms: conditions — Intervertebral disc disease

STUDY DESIGN:
Intervention Model Description: Two groups. In one the anterior annulus will be removed to insert a lumbar disc prosthesis and in the other this section of the anterior annulus will be opened up in two flaps hinged lateraly and replaced once the complete lumbar disc prosthesis is implanted
Who Masked: Participant
Masking Description: Patients will not be informed if the anterior annulus is removed or replaced
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Anterior annulus removal (Active Comparator): In these patients the anterior portion of the annulus fibrosus will be removed when inserting a complete lumbar disc prosthesis
  Interventions: Procedure: Anterior lumbar disc annulus removal versus replacement
- Anterior annulus replacement (Active Comparator): In these group of patients the anterior portion of the annulus fibrosus will be opened up in to flaps hinged lateraly and replaced once the complete lumbar disc prosthesis is inserted
  Interventions: Procedure: Anterior lumbar disc annulus removal versus replacement

INTERVENTIONS:
Procedure: Anterior lumbar disc annulus removal versus replacement — Owestry scale, SF12, Facet joint arthritis measured with Pathria scale, discal degeneration measured with Modic and Phirrmann scales

SUMMARY:
To implant a complete lumbar disc prosthesis removal of the anterior portion of the annulus fibrosus is required. As the anterior portion of the annulus limits the movement in extension and axial rotation, we would like to know how much increase these two disc movements and also the effect on the postoperative prevertebral scar on the reduction of these abnormal movement ranges. We also aim to see if repairing intraoperatively the anterior portion of the annulus has any advantage in the final result achieved.

DETAILED DESCRIPTION:
To implant a complete lumbar disc prosthesis removal of the anterior portion of the annulus fibrosus is required. It is known that the anterior portion of the annulus limits the movement in extension and axial rotation, so removal of this section of the annulus fibrosus will increase the range of movement in extension and axial rotation. As far as the investigators know, this increase in movement ranges has not been measured objectively in alive patients. Also the investigators would like to know if the postoperative prevertebral scar reduces an to what extent these abnormal movement ranges. This could help the investigators to decide when patients should be allowed to regain normal activities and specially, when the patients should be allowed to start working again. The investigators also aim to see if repairing intraoperatively the anterior portion of the annulus has any advantage in the final result achieved, and thus represents an improvement or not in the care of these patients

ELIGIBILITY:
Inclusion Criteria:

* Minimum age of 18 years and maximum of 50 years, given that above that age there is usually degenerative pathology of the lumbar joint facets, which can confuse the symptoms and make it difficult to interpret the results.
* Pathology compatible with chronic low back pain accompanied or not by radiculopathy originating in one or a maximum of two degenerated intervertebral discs and without signs of degeneration / osteoarthritis of the lumbar joint facets.
* The type of lumbar pain must be discogenic, that is, worsen in flexion and not in extension, and in loading, as well as having a truncal distribution with possible anterior radiation towards the English or genital region.
* Radiological confirmation by lumbar MRI study of lumbar discopathy of one or a maximum of two lumbar levels.
* Absence in simple radiology studies of signs of vertebral instability or listhesis of the levels to be treated.
* Absence of response for 6 weeks to conservative, non-surgical treatment, or presence of progressive symptoms. The treatment would also be carried out despite the absence of this study and the existence of the study does not condition in any way the treatment of the patients
* Not having undergone any prior treatment of the type of microdiscectomy, laminectomy or lumbar arthrodesis, although these have been carried out at different levels than those involved on this occasion
* Ability of the patient to comply with the proposed monitoring program
* Patient's ability to follow the postoperative care program
* Granting of informed consent

Exclusion Criteria:

* Signs of arthropathy of the lumbar joint facets, osteoporosis, previous interventions on the lumbar spine
* Deformity or instability of the lumbar spine
* Lumbar canal stenosis
* Previous intervention on lumbar spine
* Previous lumbar spinal fracture
* Mobile spondylolisthesis> 2 mm in translation and / or more than 11 ° angular difference with respect to the adjacent level on neutral vertical or flexion-extension radiographs
* Severe osteoporosis
* Spinal metastasis
* Metabolic bone disease that could interfere with the implant or the surgical procedure
* Rheumatoid arthritis, lupus, or other autoimmune disease that affects the musculoskeletal system
* Other conditions or anatomical alterations that make the treatment of the anterior approach to the lumbar spine unfeasible
* Known allergy to stainless steel, titanium or their alloys
* Fixed or permanent neurological deficit
* Active systemic infection at any time or ongoing preventive treatment for it, infection in the surgical site, HIV or hepatitis C
* Abusive drug or alcohol use
* Uncontrolled seizure disorder
* Psychiatric illness that could interfere with your participation in the study
* Participation in a current research study or in the 3 months prior to surgery
* History of malignancy or current malignancy (except non-melanoma skin cancer), unless the patient has been treated for curative purposes and no clinical signs or symptoms have been observed for at least 5 years
* Obesity (Body Mass Index or BMI> 35)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-28 (Estimated)

PRIMARY OUTCOMES:
Range of spinal segment movement after lumbar disc prosthesis insertion in L4-L5 lumbar disc | One year
  The investigators will analyze preoperatively and postoperatively at 3, 6 and 12 months the range of movement of the L4-L5 lumbar disc after insertion of a complete lumbar disc prosthesis

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital General Universitario de Valencia, Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Frelinghuysen P, Huang RC, Girardi FP, Cammisa FP Jr. Lumbar total disc replacement part I: rationale, biomechanics, and implant types. Orthop Clin North Am. 2005 Jul;36(3):293-9. doi: 10.1016/j.ocl.2005.02.014. PMID 15950689
- [Background] Auerbach JD, Jones KJ, Milby AH, Anakwenze OA, Balderston RA. Segmental contribution toward total lumbar range of motion in disc replacement and fusions: a comparison of operative and adjacent levels. Spine (Phila Pa 1976). 2009 Nov 1;34(23):2510-7. doi: 10.1097/BRS.0b013e3181af2622. PMID 19927100
- [Background] Huang YJ, Zhao SJ, Zhang Q, Nong LM, Xu NW. Comparison of lumbar pedicular dynamic stabilisation systems versus fusion for the treatment of lumbar degenerative disc disease: A meta-analysis. Acta Orthop Belg. 2017 Mar;83(1):180-193. PMID 29322911